CLINICAL TRIAL: NCT03439501
Title: A Phase II Study of Avelumab in Relapsed or Refractory Extranodal Natural Killer/T-cell Lymphoma
Brief Title: Avelumab in Relapsed or Refractory Extranodal Natural Killer/T-cell Lymphoma[AVENT STUDY]
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Principal Investigator, Won Seog Kim, Clinical Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-05-046; MS100070_0018 (Other Grant/Funding Number: Merck KGaA)
Record Dates: First submitted 2018-01-17; First posted 2018-02-20 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Lymphoma, Extranodal NK-T-Cell
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- avelumab (Other): * 1 Cycle: 10mg/kg Avelumab administered via IV every 2 weeks (1st, 15th)
    * Interval of 1 cycle: 28 days ③ Administration schedule: Repeated until disease progression or unacceptable toxicity and dose adjustments may be permitted based on the toxicity that occurs every cycle.
  Interventions: Drug: avelumab

INTERVENTIONS:
Drug: avelumab — * Study drug: Avelumab (PD-L1 inhibitor; MSB0010718C)
  * Dosage: 10 mg per body weight (kg) of a subject every two weeks
  * One cycle consists of two injection of avelumab (28 days).
  * The treatment cycle will be repeated until progression of disease or unacceptable toxicity and dose adjustments are permitted for patients who are unable to tolerate the side effects of drugs within each cycle.

SUMMARY:
This study was conducted to evaluate the complete response rate of avelumab in patients with NK / T-cell lymphoma besides relapsed or refractory stage lymphoma.

DETAILED DESCRIPTION:
Extranodal natural killer/T-cell lymphoma (ENKTL) generally has poorer prognosis than other lymphomas because the majority of patients are present as advanced disease and show poor response to treatment.

In particular, treatment of relapsed or refractory stage ENKTL is very poor and there is no standard treatment.

ENKTL is entirely infected with Epstein-Barr virus (EBV) and the prevalence of this disease is closely related to EBV.

Therefore, the biological properties of ENKTL may be affected by EBV-related protein and LMP1 may induce activation of molecules in various sub-channels, such as PI3K/Akt and NF-kB, and affect the aggressiveness of lymphoma.

As an increase in PDL1 has been reported recently among the major roles of LMP1, the role of Immuno-oncology drug targeting PDL1 among ENKTL is expected.

Therefore, Avelumab that inhibits PDL1 may effectively treat NK/T-cell lymphoma besides relapsed or refractory stage lymphoma.

ELIGIBILITY:
INCLUSION CRITERIA

1. Historologically diagnosed ENKTL: The standards of WHO Classification 2016 for diagnosis of ENKTL satisfied.
2. Became relapsed or refractory after at least one kind of treatment after initial diagnosis.
3. If there is at least one measurable lesion.
4. In case full-body activity (ECOG PS) is levels 0-2.
5. In case of written consent to participation in clinical study: Must sign the subject consent form that states the sampling done at the time of diagnosis or relapse (must provide sample): 10 4um (at least 5) and biomarker (3~5 ml peripheral blood drawn during screening period, must provide sample) and that the subject has comprehended the purpose and the necessary procedures of clinical study with intention to participate in the clinical study (or signed by the subject's representative).
6. If older than 19 years of age.
7. If the following hematological results are satisfied:

   * Absolute neutrophil count is 1500/mm3 or greater regardless of growth factor supply.
   * Platelet count is 100,000/mm3 or greater regardless of blood supply. (However, in cases of disease involvement, for example, platelet decrease due to bone marrow involvement or spleen enlargement, patients with a platelet count greater than 50000/mm3 may participate in this study.)
   * Hemoglobin is 9.0 g/dL or greater.
8. If the following biochemical results are satisfied:

   * Alanine transaminase (ALT) and Aspartate transaminase (AST) ≤ 2.5 x upper limit (ULN): If liver blood enzyme count is increasing due to a disease, such as the lymphoma's hepatic intrusion, may register up to ≤ 5 x ULN at investigator's discretion.
   * If bilirubin is increasing due to the Gilbert Syndrome, total bilirubin ≤ 1.5 x ULN unless non-hepatic.
   * Serum creatinine ≤ 2 x ULN or glomerular filtration rate (Cockroft Gault) ≥ 30 mL/min/1.73m2.
9. Highly efficient birth control that meets the local regulations must be adopted for birth control of subjects that participate in the clinical study during or after the clinical study for women in fertility or sexually active men (in case of women in fertility, effective birth control must be used during the administration of study drug and for 1 month after that and men must use it during the administration of studyt drug and for 3 months after that).
10. Women in fertility must show negative results at platelet (beta-chorionic gonadotropin) or pregnancy test by urine at screening.

EXCLUSION CRITERIA

1. If there is history of carcinomatous meningitis, symptomatic leptomeningeal diseases or evidence of secondary intrusion on the central nervous system based on CT or MRI scanning.
2. In case there are other carcinomas besides the target disease or in case of anamnesis of other malicious tumers during the past 3 years from the start of clinical study: Excluding basal cell carcinoma and cervical intraepithelial neoplasia that are appropriately treated.
3. If any toxicity from the previous chemotherapy has not recovered to grade 1 or lower at the time of screening; however hair loss and bone marrow inhibition are excluded and peripheral polyneuropathy may be registered at researcher's discretion if there is no risk of safety at Grade≤ 2.
4. In case of major operation within 4 weeks from registration for the clinical study or failure to recover from a major complication of such operation.
5. If using immunosuppressant drugs at the time of registration for the clinical study: Excluding local steroid injections such as nasal or inhalated steroid, steroid ointment, and injections in articular cavities. In case of full-body steroid administration, 10 mg or smaller prednisolonum a day is permissible (If adrenal insufficiency is necessary to maintain a dose of prednisolone 10 mg or more, it is acceptable according to the investigator's judgment) and steroid injections used for pre-treatment before CT or other examination are also permitted.
6. In case of uncontrolled or symptomatic arrhythmia, congestive heart failure, myocardial infarction, cerebral infarction, or other clinically significant cardiovascular diseases or Class 3 (Moderate) or Class 4 (Severe) cardiac diseases functionally classified by New York Heart Association within 6 months of screening.
7. In case of history of serious hypersensitivity against the study drug used for this study or its substances including serious hypersensitivity against monoclonal antibody (NCI CTCAE v4.03 Grade ≥ 3).
8. In case of known history of human immunodeficiency virus (HIV), active type C hepatitis virus, or active type B hepatitis virus (However, in the case of healthy carriers who did not require asymptomatic treatment, if the antiviral drug can be taken, it can be registered by the judgment of the investigator. In this case, the HBV DNA test should be monitored periodically through division of gastroenterology) or uncontrolled active full-body infection that requires intravenous (IV) antibiotics.
9. In case of life-threatening diseases, medical conditions, or respiratory failure that may threaten the safety of subjects or put the results of clinical study in danger.
10. In case of homogeneous hematopoietic stem cell transplant.
11. In case of active autoimmune disease that may affect the administration of study drug; excluding type 1diabetes, psoriasis, vitiligo, hyperthyroidism, or hypothyroidism that does not require immunosuppressant.
12. If the candidate cannot comprehend the clinical study or comply with the rules of clinical study including an active attempt to commit suicide or hurt oneself recently or in the past and other severe acute or chronic diseases such as immunocolitis, ulcerative colitis, immunopneumonia, pulmonary fibrosis, or mental conditions; or if determined by investigator that participation in the study is inappropriate due to any risk of participation or treatment in the study that may increase due to adverse effects or the interpretation of study results that may be hindered.
13. If candidate is pregnant or breast-feeding at the time of screening.
14. In case of a major operation or live attenuated vaccine within 4 weeks of registration for the clinical study.
15. In case of the following hepatic diseases:

    * Chronic hepatitis or liver cirrhosis related to type B or type C hepatitis.
    * Positive reaction for surface antigen of type B hepatitis without symptoms. (However, in the case of healthy carriers who did not require asymptomatic treatment, if the antiviral drug can be taken, it can be registered by the judgment of the investigator. In this case, the HBV DNA test should be monitored periodically through division of gastroenterology): Positive reaction to RNA of type C hepatitis without symptoms.
16. Previously exposed to PD-1 / PD-L1 inhibitor
17. Use of other anticancer treatment or other study drugs within 4 weeks of registration for the clinical study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
The rate of response of avelumab. | From date of enrollment until the date first documented disease progression or unacceptable toxicity, whichever came first, assessed up to 48 months
  To assess the efficacy of disease control including complete response (CR), partial response (PR) and stable disease (SD)

SECONDARY OUTCOMES:
Progression-free survival | the time between the date of treatment start and the date of death due to any cause or date of disease progression..assessed up to 48 months
  It is a measure of the period of survival without disease progression
Overall survival (OS) | Time between the start of treatment and the date of death.assessed up to 48 months
  It measures the time from start of treatment to death.
Toxicity Profile | from the date of informed consent signature to 30 days after last drug administration.
  Clinical and laboratory toxicity/symptomatology will be graded based on the NCIC CTG v4.03. Adverse events not reported in NCIC CTG will be categorized into mild, moderate, severe, and fatal and further classified to CTCAE Grades 1-4.

CONTACTS AND LOCATIONS:
Overall Officials: Wonseog Kim, M.D, Principal Investigator — Samsung Medical Center
Locations (1):
- 81, Irwon-ro, Gangnam-gu, Seoul, Republic of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim SJ, Lim JQ, Laurensia Y, Cho J, Yoon SE, Lee JY, Ryu KJ, Ko YH, Koh Y, Cho D, Lim ST, Enemark MB, D'Amore F, Bjerre M, Ong CK, Kim WS. Avelumab for the treatment of relapsed or refractory extranodal NK/T-cell lymphoma: an open-label phase 2 study. Blood. 2020 Dec 10;136(24):2754-2763. doi: 10.1182/blood.2020007247. PMID 32766875